CLINICAL TRIAL: NCT02752425
Title: Visual Feedback of Tongue by Ultrasound Echography for Speech Trouble Rehabilitation
Acronym: REVISON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL15_0736
Record Dates: First submitted 2016-04-21; First posted 2016-04-27 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2019-01

CONDITIONS: Speech Disorders
Keywords: Speech disorders; Speech therapy; Visual feedback; Buccopharyngeal surgery; Central nervous system damage
MeSH Terms: conditions — Speech Disorders; Communication Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With visual feedback (Experimental): Session of speech therapy conducted with the additional use of articulatory visual feedback based on ultrasound echography, which allows to visualize the patient's tongue in real time on a computer screen
  Interventions: Device: Visual feedback
- Without visual feedback (No Intervention): Session of speech therapy without use of ultrasound echography

INTERVENTIONS:
Device: Visual feedback — Use of ultrasound echography for tongue articulatory visual feedback
  Arms: With visual feedback

SUMMARY:
Speech is a privileged means of communication for humans: its trouble can thus prove being extremely handicapping. Standard speech therapy is limited in some cases by the lack of sensory feedback available to the patient (hearing, surgery, neural damage, etc.).

The present study aims at quantify the contribution of the tongue articulatory visual feedback offered by ultrasound echography to speech trouble rehabilitation.

Two complementary populations will be studied : 30 adults with buccopharyngeal surgery, and 10 childrens with important speech troubles due to central nervous system damage.

The principle is to conduct standard speech therapy sessions, alternating series of sessions with the use of visual feedback and sessions without visual feedback.

The progress will be regularly measured by means of standard batteries of speech articulation tests.

ELIGIBILITY:
Inclusion Criteria:

* Articulatory troubles needing speech therapy
* French mother tongue
* Adult patients [18 ≥ age < 80 years] who underwent buccopharyngeal surgery after cancer diagnostic OR children [8 ≥ age < 18 years] suffering from central nervous system damage

Exclusion Criteria:

* Incapacity to easily understand the speech therapist instructions
* People protected by the law
* People deprived from freedom by judiciary decision
* Potential allergy to the water-based conducting gel used to ensure good skin - probe contact
* Overweight if large fatty mass under chin
* Major edema under chin limiting echogenicity
* Non corrected vision or hearing problems
* For the adults: central or peripheral neural damage
* History of Ear, Nose, and Throat surgery or radiotherapy
* For the adults: isolated articulatory trouble, former articulatory trouble not treated, disfluency
* Massive orofacial dyspraxia
* Posture trouble
* Motor problem in upper limbs

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
BECD test score | 4 months
  One of the primary outcome will be measured as the difference of increase of total BECD score between the therapy sessions with and without visual feedback.
  BECD ("Batterie d'Evaluation Clinique de la Dysarthrie, Battery of Clinical Evaluation of Dysarthria") is a French speech articulation test.
MBLF test score | 4 months
  The second primary outcome will be measured as the difference of increase of total MBLF score between the therapy sessions with and without visual feedback.
  MBLF ("Motricité Bucco-Linguo-Faciale, Motricity of Mouth, Tongue and Face") is a French speech articulation test.

SECONDARY OUTCOMES:
Perception test scores | 4 months
  The secondary outcome will be measured as the difference of increase of the scores of perception obtained by a jury listening to a selected set of patients' speech sounds between the therapy sessions with and without visual feedback. The speech sounds are those recorded during the batteries of speech articulation tests.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BADIN, PhD, Study Director — GIPSA-lab, CNRS, Univ. Grenoble Alpes
Locations (2):
- France (2):
  - Institut d'Education Motrice, Eybens
  - Centre Médical Rocheplane, Saint-Martin-d'Hères

REFERENCES:
- [Result] Girod-Roux M, Hueber T, Fabre D, Gerber S, Canault M, Bedoin N, Acher A, Beziaud N, Truy E, Badin P. Rehabilitation of speech disorders following glossectomy, based on ultrasound visual illustration and feedback. Clin Linguist Phon. 2020 Sep 1;34(9):826-843. doi: 10.1080/02699206.2019.1700310. Epub 2020 Jan 28. PMID 31992079